CLINICAL TRIAL: NCT02576548
Title: A Phase 1/2 Multicenter, Open-label, Dose-escalation, and Dose-expansion Study to Evaluate the Safety, Pharmacokinetics, Immunogencity, and Antitumor Activity of MEDI4276 in Subjects With Select HER2-expressing Advanced Solid Tumors
Brief Title: A Phase 1/2 Study of MEDI4276 in Adults Subjects With Select HER2-expressing Advanced Solid Tumors.
Acronym: MEDI4276
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5760C00001
Record Dates: First submitted 2015-09-28; First posted 2015-10-15 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: HER2 Expressing Breast or Gastric/Stomach Cancers
MeSH Terms: conditions — Stomach Neoplasms | interventions — MEDI4276

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- MEDI4276 0.05 mg/kg (Experimental): Participants received IV dose of 0.05 mg/kg MEDI4276 every three weeks (Q3W) for 2 years.
  Interventions: Biological: MEDI4276
- MEDI4276 0.1 mg/kg (Experimental): Participants received IV dose of 0.1 mg/kg MEDI4276 every three weeks (Q3W) for 2 years.
  Interventions: Biological: MEDI4276
- MEDI4276 0.2 mg/kg (Experimental): Participants received IV dose of 0.2 mg/kg MEDI4276 every three weeks (Q3W) for 2 years.
  Interventions: Biological: MEDI4276
- MEDI4276 0.3 mg/kg (Experimental): Participants received IV dose of 0.3 mg/kg MEDI4276 every three weeks (Q3W) for 2 years.
  Interventions: Biological: MEDI4276
- MEDI4276 0.4 mg/kg (Experimental): Participants received IV dose of 0.4 mg/kg MEDI4276 every three weeks (Q3W) for 2 years.
  Interventions: Biological: MEDI4276
- MEDI4276 0.5 mg/kg (Experimental): Participants received IV dose of 0.5 mg/kg MEDI4276 every three weeks (Q3W) for 2 years.
  Interventions: Biological: MEDI4276
- MEDI4276 0.6 mg/kg (Experimental): Participants received IV dose of 0.6 mg/kg MEDI4276 every three weeks (Q3W) for 2 years.
  Interventions: Biological: MEDI4276
- MEDI4276 0.75 mg/kg (Experimental): Participants received IV dose of 0.75 mg/kg MEDI4276 every three weeks (Q3W) for 2 years.
  Interventions: Biological: MEDI4276
- MEDI4276 0.9 mg/kg (Experimental): Participants received IV dose of 0.9 mg/kg MEDI4276 every three weeks (Q3W) for 2 years.
  Interventions: Biological: MEDI4276

INTERVENTIONS:
Biological: MEDI4276 — MEDI4276 is an investigational product

SUMMARY:
This research study is designed to evaluate an experimental drug, MEDI4276, in treating breast and stomach (gastric) cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histologically or cytologically documented unresectable, locally advanced or metastatic breast cancer or gastric cancer refractory to standard therapy.

   1. For subjects with breast cancer:

      * Prior treatment with trastuzumab, pertuzumab, and T-DM1, either alone or in combination, is required.
      * Subjects with a primary tumor that is hormone (estrogen, progesterone, or both) receptor-positive or receptor-negative are eligible.
      * Prior hormone therapy is allowed, but last dose must be at least 14 days prior to first dose of MEDI4276.
   2. For subjects with gastric cancer:

      * Prior treatment with a trastuzumab containing chemotherapy regimen is required.
3. HER2 Positive disease documented as FISH-positive and/or 3+ by IHC on previously collected tumor tissue.
4. At least one lesion measurable by RECIST Version 1.1.

Exclusion Criteria:

1. Receipt of any conventional or investigational anticancer treatment within 28 days prior to the first dose of MEDI4276.
2. History of exposure to the following cumulative doses of anthracyclines:

   1. Doxorubicin or liposomal doxorubicin >350 mg/m².
   2. Epirubicin >530 mg/m².
   3. Mitoxantrone >90 mg/m² and idarubicin > 70 mg/m².
   4. If another anthracycline or more than 1 anthracycline has been used, then the cumulative dose must not exceed the equivalent of 350 mg/m² of doxorubicin.
3. Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms; or any radiation, surgery or other therapy to control symptoms from brain metastases within 2 months prior to first dose of MEDI4276.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Number and percentage of subjects with adverse events (AEs), serious adverse events (SAEs) and dose-limiting (DLTs). | From Time of informed consent through 90 days after last dose of MEDI4276
  The maximum tolerated dose/maximum administered dose will be determined by the number of participants experiencing DLTs. The safety profile will be assessed through number of participants experiencing AEs, SAEs, abnormal laboratory parameters, vital signs and electrocardiogram (ECG) results.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Time from Informed Consent up to 3 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR
Peak Plasma Concentration (Cmax) | From first dose of MEDI4276 thorugh to 30 days after last dose of investigational product
  The immunogenicity of MEDI4276 will be assessed by summarizing the number and percentage of subjects who develop detectable anti-drug antibodies (ADAs)
Progression-free survival (PFS) | Estimated to be from time of informed consent up to 3 years
  Progression-free survival will be measured from the start of treatment with MEDI4276 until the first documentation of confirmed immune-related disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Estimated to be from time of informed consent up to 3 years
  Overall survival will be determined as the time from the start of treatment with MEDI4276 until death due to any cause.
Area under the plasma concentration versus time curve (AUC) | From first dose of MEDI4276 through to 30 days after the last dose of investigational product
  The immunogencity of MEDI 4276 will be assessed by summarizing the number and percentage of subjects who develop detectable anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — Sponsor GmbH
Locations (5):
- United States (5):
  - Research Site, Stanford, California
  - Research Site, Sarasota, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Charlotte, North Carolina
  - Research Site, Nashville, Tennessee

REFERENCES:
- [Derived] Faria M, Peay M, Lam B, Ma E, Yuan M, Waldron M, Mylott WR Jr, Liang M, Rosenbaum AI. Multiplex LC-MS/MS Assays for Clinical Bioanalysis of MEDI4276, an Antibody-Drug Conjugate of Tubulysin Analogue Attached via Cleavable Linker to a Biparatopic Humanized Antibody against HER-2. Antibodies (Basel). 2019 Jan 11;8(1):11. doi: 10.3390/antib8010011. PMID 31544817